CLINICAL TRIAL: NCT06865612
Title: Optimizing Accuracy: a Comparative Analysis of Preoperative Liver Volumetry in Living Donor Liver Transplantation from a Surgeon's Perspective
Brief Title: A Comparative Analysis of Preoperative Liver Volumetry in Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-05-025
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Living Donor Liver Transplantation; Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Donors: Patients who received hepatectomy for the living donor liver transplantation.

SUMMARY:
Accurate preoperative graft volume assessment is crucial for successful living donor liver transplantation (LDLT). Although manual and automated computed tomography (CT) volume measurement methods using various volumetric tools are widely used, their accuracy remains uncertain. This study aimed to determine the optimal dry weight correction factor for each method to enhance the prediction of actual graft weight (AGW) and compare the accuracy of different methods.

DETAILED DESCRIPTION:
This study is a retrospective diagnostic accuracy study comparing three liver volumetry methods using preoperative donor CT scans in LDLT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent hepatectomy for living donor liver transplantation performed by the Department of Surgery at Chungnam National University Hospital under the supervision of the principal investigator.

Exclusion Criteria:

* Patients deemed unsuitable for participation in this clinical study by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients who underwent hepatectomy for living donor liver transplantation performed at Chungnam National University Hospital. Data will be retrospectively reviewed to compare preoperative estimated graft volume (EGV) to actual graft weight (AGW).
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of preoperative estimated graft volume (EGV) compared to actual graft weight (AGW) | From preoperative CT scan (1-2 months before transplantation) to intraoperative measurement (day of transplantation)
  The accuracy of preoperative donor CT liver volumetry will be assessed by comparing estimated graft volume (EGV) obtained from three methods (automated, semi-automated, manual) with the actual graft weight (AGW) measured intraoperatively. The error ratio between EGV and AGW will be calculated for each method.

SECONDARY OUTCOMES:
Determination of the optimal dry weight correction factor for each volumetry method | From preoperative CT scan (1-2 months before transplantation) to intraoperative measurement (day of transplantation)
  The study aims to determine the optimal dry weight correction factor by minimizing the discrepancy between EGV and AGW.

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No
The data will not be shared publicly due to the retrospective nature of the study and privacy protection concerns.